CLINICAL TRIAL: NCT03894618
Title: Phase 1 Dose Escalation and Dose Expansion Study of an Agonist Redirected Checkpoint Fusion Protein, SL-279252 (PD1-Fc-OX40L), in Subjects With Advanced Solid Tumors or Lymphomas
Brief Title: SL-279252 (PD1-Fc-OX40L) in Subjects With Advanced Solid Tumors or Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shattuck Labs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SL01-DEL-101
Record Dates: First submitted 2019-01-10; First posted 2019-03-28 (Actual); Results first posted 2025-03-14 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-02

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck; Melanoma; Non Small Cell Lung Cancer; Urothelial Carcinoma; Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma; Squamous Cell Carcinoma of the Anus; Squamous Cell Carcinoma of the Cervix; Squamous Cell Carcinoma of the Skin; Renal Cell Carcinoma; Hodgkin Lymphoma; Diffuse Large B Cell Lymphoma; Mismatch Repair Deficient or MSI-High Solid Tumors
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Melanoma; Carcinoma, Non-Small-Cell Lung; Carcinoma, Transitional Cell; Anus Neoplasms; Carcinoma, Renal Cell; Hodgkin Disease; Lymphoma, Large B-Cell, Diffuse; Turcot syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SL-279252 (Experimental): Intravenous administration; Two possible dosing schedules for SL-279252 may be evaluated
  Interventions: Drug: SL-279252

INTERVENTIONS:
Drug: SL-279252 — The investigational product (IP), SL-279252, is a first-in-class agonist redirected checkpoint (ARC) fusion protein (FP) consisting of the extracellular domains of human programmed cell death 1 (PD- 1) and OX40L, linked by a central Fc domain (PD1-Fc-OX40L).

SUMMARY:
This is a Phase 1 first in human, open label, multi-center, dose escalation and dose expansion study to evaluate the safety, tolerability, PK, anti-tumor activity and pharmacodynamic effects of SL-279252 in subjects with advanced solid tumors or lymphomas.

DETAILED DESCRIPTION:
This is a Phase 1 first in human, open label, multi-center, dose escalation and dose expansion study to evaluate the safety, tolerability, PK, anti-tumor activity and pharmacodynamic effects of SL-279252 in subjects with advanced solid tumors or lymphomas. The study design consists of Dose Escalation and Dose Expansion Cohorts. In the dose escalation phase of the study, subjects will be enrolled into sequential dose levels. During dose escalation, two possible schedules for administration of SL-279252 may be explored. The MTD or MAD may be determined for either schedule. Based on accumulating data from the dose escalation phase, including safety, PK, pharmacodynamic and anti-tumor activity, up to two dose expansion cohorts may be opened. The primary objective of the expansion phase is to further refine the safety and tolerability of SL-279252. The expansion cohorts will evaluate one or two doses of SL-279252 using one selected schedule. At the end of dose escalation and dose expansion, safety, PK, anti-tumor activity, and pharmacodynamic data will be reviewed to identify the RP2D.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all the following criteria apply.

1. Subject has voluntarily agreed to participate by giving written informed consent in accordance with ICH/GCP guidelines and applicable local regulations.
2. Subject has a histologically confirmed diagnosis of one of the following unresectable locally advanced or metastatic malignancies: melanoma, non-small cell lung cancer (squamous, adeno, or adeno-squamous), urothelial cancer, squamous cell carcinoma of the head and neck, squamous cell cervical cancer, gastric or gastro-esophageal junction adenocarcinoma, squamous cell carcinoma of the anal canal, squamous cell carcinoma of the skin, renal cell cancer, Hodgkin's lymphoma, and microsatellite instability high (MSI-H) or mismatch repair deficient (MMRD) solid tumors excluding CNS malignancies. MSI and MMRD testing results as per institution is acceptable.

   * Head and neck cancers: Subjects must have primary tumor locations in the oropharynx, oral cavity, hypopharynx, or larynx. Primary tumor sites of nasopharynx, maxillary sinus, paranasal, and unknown primary are excluded.
   * Non-small cell lung cancers: Subjects with a known EGFR sensitizing (activating) mutation or an ALK fusion are excluded.
3. Subject must have received, been intolerant to, or is ineligible for standard therapy (per local guidelines and approvals) or have a malignancy for which there is no approved therapy considered standard of care.
4. Age 18 years and older.
5. Has an Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1.
6. Has measurable disease by iRECIST (solid tumors) or RECIL 2017 (lymphoma). Refer to Appendix Sections 16.6 and 16.7 for details on criteria of measurable disease.
7. Has life expectancy of greater than 12 weeks.
8. Laboratory values must meet the following criteria. Laboratory parameter Threshold value

   * Absolute lymphocyte count (ALC) ≥ 0.8 x 109/liter (L)
   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L without growth factor support
   * Platelet count ≥ 50 x 109/L

   Laboratory parameter Threshold value
   * Hemoglobin (Hgb) > 9.0 g/dL with no blood transfusions for at least 5 days prior to D1 of investigational product (IP; SL-279252)
   * Creatinine clearance (CrCl) ≥ 30 milliliter (mL)/min (modified Cockcroft-Gault)
   * ALT/AST ≤ 3 x ULN
   * Total bilirubin ≤ 1.5 x ULN; subjects with isolated indirect hyperbilirubinemia are permitted if direct bilirubin ratio is <35% and total bilirubin is ≤ 3.0 x ULN
   * Left ventricular ejection fraction (LVEF) by echocardiogram (ECHO) ≥ lower limit of normal (LLN) per institutional threshold. If LLN is not defined for a given institution, then ejection fraction must be ≥50 %.
9. Females of child bearing potential (FCBP) must have a negative serum or urine pregnancy test within 72 hours of D1 of IP. NOTE: FCBP unless they are surgically sterile (i.e., have undergone a complete hysterectomy, bilateral tubal ligation/occlusion, bilateral oophorectomy or bilateral salpingectomy), have a congenital or acquired condition that prevents childbearing or are naturally postmenopausal for at least 12 consecutive months (see Appendix Section 16.2 for additional details). Documentation of postmenopausal status must be provided. FCBP should use an acceptable method of contraception (see Appendix Section 16.2) to avoid pregnancy during treatment and for 30 days (which exceeds 5 half-lives) after the last dose of IP. FCBP must start using acceptable contraception at least 14 days prior to D1 of IP.
10. Male subjects with female partners must have azoospermia from a prior vasectomy or underlying medical condition or agree to use an acceptable method of contraception during treatment and for 30 days (which exceeds 5 half-lives) after last dose of SL-279252 (see Appendix Section 16.2). Male subjects of reproductive potential must start using acceptable contraception at least 14 days prior to D1 of treatment with SL-279252 as per Appendix Section 16.2.
11. All AEs resulting from prior anti-cancer immunotherapy have resolved (NOTE: exceptions include alopecia, vitiligo, and endocrinopathies adequately treated with hormone replacement).

    • Subjects that were discontinued from prior PD-1/L1 therapy due to immune-related adverse events are not eligible
12. Recovery from toxicities from prior anti-cancer treatments including surgery, radiotherapy, chemotherapy or any other anti-cancer therapy to baseline or ≤ Grade 1. (NOTE: Low-grade toxicities (e.g., alopecia, ≤ Grade 2 lymphopenia, ≤ Grade 2 hypomagnesemia, ≤ Grade 2 neuropathy) may be allowed at the discretion of the investigator if considered clinically insignificant. Please consult the Sponsor Medical Monitor to discuss these cases).

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. Has received more than two prior checkpoint inhibitor containing treatment regimens (regimen refers to either monotherapy or combination immunotherapies) or has had prior treatment with an OX40 agonist.

   • Prior PD-1/L1 therapy is not required.
2. Refractory to last PD-1/L1 inhibitor-based therapy which is defined as disease progression within 3 months of treatment initiation.

   • Subjects must have had clinical benefit (stable disease or response) to last PD-1/L1 inhibitor-based therapy for at least three months to be eligible.
3. Any anti-cancer therapy within the time intervals noted below prior to first dose (D1) of SL-279252.

   Therapy Washout period Chemotherapy 3 weeks Hormonal therapy 3 weeks PD-1/L1 inhibitor and other immunotherapies not otherwise specified 3 weeks Tumor vaccine 4 weeks Cell-based therapy 8 weeks Other mAbs or biologic therapies 3 weeks Major surgery 2 weeks Radiation (except palliative intent which does not require washout) 2 weeks
4. Concurrent chemotherapy, immunotherapy, biologic or hormonal therapy is prohibited. Concurrent use of hormones for non-cancer related conditions is acceptable.
5. Use of corticosteroids or other immunosuppressive medication, current or within 14 days of D1 of IP with the following exceptions (i.e., the following are allowed during treatment with or within14 days of D1 of IP):

   * Topical, intranasal, inhaled, ocular, intraarticular corticosteroids
   * Physiological doses of replacement steroid (e.g., for adrenal insufficiency) provided ≤ 10 mg/day of prednisone or equivalent
   * Steroid premedication for hypersensitivity reactions (HSRs; e.g., reaction to IV contrast)
6. Receipt of live attenuated vaccine within 28 days of D1 of IP.
7. Active or documented history of autoimmune disease (autoimmune disease does not refer to irAEs; for irAEs see inclusion criteria #11). Exceptions include Type I diabetes, vitiligo, alopecia areata or hypo/hyperthyroidism.
8. Active pneumonitis (i.e. drug-induced, idiopathic pulmonary fibrosis, radiation-induced, etc.).
9. Ongoing or active infection (e.g., no systemic antimicrobial therapy for treatment of infection within 5 days of D1 of IP).
10. Symptomatic peptic ulcer disease or gastritis, active diverticulitis, other serious gastrointestinal (GI) disease associated with diarrhea within 6 months of D1 of IP.
11. Clinically significant or uncontrolled cardiac disease including any of the following:

    * Myocarditis
    * Unstable angina within 6 months from D1 of IP
    * Acute myocardial infarction within 6 months from D1 of IP
    * Uncontrolled hypertension
    * New York Heart Association (NYHA) Class II, III or IV congestive heart failure
    * Clinically significant (symptomatic) cardiac arrhythmias (e.g., sustained ventricular tachycardia, second- or third- degree atrioventricular block without a pacemaker, circulatory collapse requiring vasopressor or inotropic support, or arrhythmia requiring therapy)
12. Untreated central nervous system (CNS) or leptomeningeal metastases. Subjects with treated CNS metastases must have completed definitive treatment (radiotherapy and/or surgery) > 2 weeks prior to D1 of IP and no longer require steroids.
13. Women who are breast feeding.
14. Psychiatric illness/social circumstances that would limit compliance with study requirements and substantially increase the risk of AEs or compromised ability to provide written informed consent.
15. Another malignancy that requires active therapy and that in the opinion of the investigator and Sponsor would interfere with monitoring of radiologic assessments of response to IP.
16. Has undergone allogeneic stem cell transplantation or organ transplantation.
17. Known history or positive test for human immunodeficiency virus, or positive test for hepatitis B (positive for hepatitis B surface antigen [HBsAg]) or hepatitis C virus ([HCV]; if HCV antibody (Ab) test is positive check for HCV ribonucleic acid [RNA]).

    * (NOTE: Hepatitis B virus (HBV): Subjects who are hepatitis B core antibody [HBcAb] positive, but HBsAg negative are eligible for enrollment. HCV: Subjects who are HCV Ab positive, but HCV RNA negative are eligible for enrollment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shattuck Labs, Study Director — Shattuck Labs
Locations (5):
- United States (2):
  - The Sarah Cannon Research Institute, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Leuven Cancer Institute, Leuven, Belgium
- Princess Margaret Cancer Center, Toronto, Ontario, Canada
- Vall d'Hebron Institut D' Oncologia, Barcelona, Spain

REFERENCES:
- [Derived] Johnson M, Hong D, Brana I, Schoffski P, Galvao V, Rangwala F, Ma B, Hernandez R, Kamat A, Kato K, Schreiber TH, Pandite L, Siu LL. First-in-human, phase 1 dose escalation study of SL-279252, a hexameric PD1-Fc-OX40L fusion protein, in patients with advanced solid tumors and lymphoma. Invest New Drugs. 2025 Apr;43(2):284-292. doi: 10.1007/s10637-025-01518-7. Epub 2025 Mar 5. PMID 40042547

RESULTS

PARTICIPANT FLOW:
Groups:
- SL-279252 (0.0001 mg/kg S1): 0.0001 mg/kg of IV SL-279252 (Schedule 1)
- SL-279252 (0.001 mg/kg S1): 0.001 mg/kg of IV SL-279252 (Schedule 1)
- SL-279252 (0.003 mg/kg S1): 0.003 mg/kg of IV SL-279252 (Schedule 1)
- SL-279252 (0.01 mg/kg S1): 0.01 mg/kg of IV SL-279252 (Schedule 1)
- SL-279252 (0.03 mg/kg S1): 0.03 mg/kg of IV SL-279252 (Schedule 1)
- SL-279252 (0.1 mg/kg S1): 0.1 mg/kg of IV SL-279252 (Schedule 1)
- SL-279252 (0.3 mg/kg S1): 0.3 mg/kg of IV SL-279252 (Schedule 1)
- SL-279252 (1.0 mg/kg S1): 1.0 mg/kg of IV SL-279252 (Schedule 1)
- SL-279252 (3.0 mg/kg S1): 3.0 mg/kg of IV SL-279252 (Schedule 1)
- SL-279252 (6.0 mg/kg S1): 6.0 mg/kg of IV SL-279252 (Schedule 1)
- SL-279252 (12.0 mg/kg S1): 12.0 mg/kg of IV SL-279252 (Schedule 1)
- SL-279252 (24.0 mg/kg S1): 24.0 mg/kg of IV SL-279252 (Schedule 1)
- SL-279252 (0.3 mg/kg S2): 0.3 mg/kg of IV SL-279252 (Schedule 2)
- SL-279252 (1.0 mg/kg S2): 1.0 mg/kg of IV SL-279252 (Schedule 2)
- SL-279252 (3.0 mg/kg S2): 3.0 mg/kg of IV SL-279252 (Schedule 2)
Period: Overall Study
Arm/Group | SL-279252 (0.0001 mg/kg S1) | SL-279252 (0.001 mg/kg S1) | SL-279252 (0.003 mg/kg S1) | SL-279252 (0.01 mg/kg S1) | SL-279252 (0.03 mg/kg S1) | SL-279252 (0.1 mg/kg S1) | SL-279252 (0.3 mg/kg S1) | SL-279252 (1.0 mg/kg S1) | SL-279252 (3.0 mg/kg S1) | SL-279252 (6.0 mg/kg S1) | SL-279252 (12.0 mg/kg S1) | SL-279252 (24.0 mg/kg S1) | SL-279252 (0.3 mg/kg S2) | SL-279252 (1.0 mg/kg S2) | SL-279252 (3.0 mg/kg S2)
Started | 1 | 1 | 2 | 1 | 2 | 3 | 4 | 6 | 6 | 4 | 4 | 2 | 4 | 6 | 3
Completed | 1 | 1 | 2 | 1 | 2 | 3 | 4 | 6 | 6 | 4 | 4 | 2 | 4 | 6 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SL-279252 (0.0001 mg/kg S1) | SL-279252 (0.001 mg/kg S1) | SL-279252 (0.003 mg/kg S1) | SL-279252 (0.01 mg/kg S1) | SL-279252 (0.03 mg/kg S1) | SL-279252 (0.1 mg/kg S1) | SL-279252 (0.3 mg/kg S1) | SL-279252 (1.0 mg/kg S1) | SL-279252 (3.0 mg/kg S1) | SL-279252 (6.0 mg/kg S1) | SL-279252 (12.0 mg/kg S1) | SL-279252 (24.0 mg/kg S1) | SL-279252 (0.3 mg/kg S2) | SL-279252 (1.0 mg/kg S2) | SL-279252 (3.0 mg/kg S2) | Total
Number analyzed (Participants) | 1 | 1 | 2 | 1 | 2 | 3 | 4 | 6 | 6 | 4 | 4 | 2 | 4 | 6 | 3 | 49
Age, Continuous [Median (Full Range); unit: years] | 68.0 [68 to 68] | 70.0 [70 to 70] | 51.5 [48 to 55] | 58.0 [58 to 58] | 48.5 [31 to 66] | 68.0 [63 to 77] | 74.5 [66 to 81] | 61.5 [41 to 81] | 53.0 [43 to 73] | 65.0 [50 to 66] | 65.0 [62 to 71] | 66.5 [60 to 73] | 68.5 [64 to 82] | 60.0 [38 to 70] | 62.0 [44 to 62] | 64.0 [31 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 1 | 0 | 0 | 3 | 4 | 4 | 1 | 3 | 1 | 0 | 2 | 2 | 23
  Male | 1 | 0 | 1 | 0 | 2 | 3 | 1 | 2 | 2 | 3 | 1 | 1 | 4 | 4 | 1 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 1 | 0 | 2 | 1 | 1 | 3 | 4 | 6 | 6 | 3 | 3 | 2 | 4 | 6 | 3 | 45
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  White | 1 | 1 | 1 | 0 | 2 | 3 | 4 | 6 | 6 | 4 | 2 | 2 | 4 | 6 | 2 | 44
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 1 | 0 | 2 | 3 | 1 | 2 | 3 | 1 | 4 | 1 | 3 | 0 | 0 | 23
  Canada | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 2 | 2 | 11
  Spain | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 1 | 0 | 0 | 0 | 3 | 1 | 10
  Belgium | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Safety Profile of SL-279252
Description: Number of participants with treatment emergent adverse events
Time Frame: From Day 1 to 90 days after Last Dose of SL-279252
Measure: Count of Participants; unit: Participants
Arm/Group | SL-279252 (0.0001 mg/kg S1) | SL-279252 (0.001 mg/kg S1) | SL-279252 (0.003 mg/kg S1) | SL-279252 (0.01 mg/kg S1) | SL-279252 (0.03 mg/kg S1) | SL-279252 (0.1 mg/kg S1) | SL-279252 (0.3 mg/kg S1) | SL-279252 (1.0 mg/kg S1) | SL-279252 (3.0 mg/kg S1) | SL-279252 (6.0 mg/kg S1) | SL-279252 (12.0 mg/kg S1) | SL-279252 (24.0 mg/kg S1) | SL-279252 (0.3 mg/kg S2) | SL-279252 (1.0 mg/kg S2) | SL-279252 (3.0 mg/kg S2)
Number analyzed (Participants) | 1 | 1 | 2 | 1 | 2 | 3 | 4 | 6 | 6 | 4 | 4 | 2 | 4 | 6 | 3
Participants | 1 | 1 | 2 | 1 | 2 | 3 | 4 | 5 | 6 | 3 | 4 | 2 | 4 | 5 | 3

2. Primary Outcome: Maximum Tolerated Dose (MTD) of SL-279252
Description: Number of participants with dose limiting toxicities (DLTs)
Time Frame: From Day 1 to Day 21 (Schedule 1) or Day 28 (Schedule 2)
Population: DLT evaluable population
Measure: Count of Participants; unit: Participants
Arm/Group | SL-279252 (0.0001 mg/kg S1) | SL-279252 (0.001 mg/kg S1) | SL-279252 (0.003 mg/kg S1) | SL-279252 (0.01 mg/kg S1) | SL-279252 (0.03 mg/kg S1) | SL-279252 (0.1 mg/kg S1) | SL-279252 (0.3 mg/kg S1) | SL-279252 (1.0 mg/kg S1) | SL-279252 (3.0 mg/kg S1) | SL-279252 (6.0 mg/kg S1) | SL-279252 (12.0 mg/kg S1) | SL-279252 (24.0 mg/kg S1) | SL-279252 (0.3 mg/kg S2) | SL-279252 (1.0 mg/kg S2) | SL-279252 (3.0 mg/kg S2)
Number analyzed (Participants) | 1 | 1 | 2 | 1 | 2 | 3 | 4 | 3 | 5 | 3 | 4 | 2 | 3 | 6 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Recommended Phase 2 Dose for SL-279252
Description: Based on review of all data, including safety, tolerability, PK, antitumor activity, and PD effects
Time Frame: Approximately 32 months
Measure: Number; unit: mg/kg
Groups:
- SL-279252: SL-279252 received in Schedule 1 or Schedule 2
Arm/Group | SL-279252
Number analyzed (Participants) | 49
mg/kg | NA — MTD/RP2D not achieved in this study

4. Secondary Outcome: Overall Response Rate of SL-279252
Description: Objective response rate per immune response evaluation criteria in solid tumors (iRECIST) for solid tumors
Time Frame: Approximately 32 months
Population: All treated population with solid tumors
Measure: Count of Participants; unit: Participants
Arm/Group | SL-279252 (0.0001 mg/kg S1) | SL-279252 (0.001 mg/kg S1) | SL-279252 (0.003 mg/kg S1) | SL-279252 (0.01 mg/kg S1) | SL-279252 (0.03 mg/kg S1) | SL-279252 (0.1 mg/kg S1) | SL-279252 (0.3 mg/kg S1) | SL-279252 (1.0 mg/kg S1) | SL-279252 (3.0 mg/kg S1) | SL-279252 (6.0 mg/kg S1) | SL-279252 (12.0 mg/kg S1) | SL-279252 (24.0 mg/kg S1) | SL-279252 (0.3 mg/kg S2) | SL-279252 (1.0 mg/kg S2) | SL-279252 (3.0 mg/kg S2)
Number analyzed (Participants) | 1 | 1 | 2 | 1 | 2 | 3 | 4 | 5 | 6 | 4 | 4 | 2 | 4 | 6 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Immunogenicity to SL-279252
Description: Number of participants with positive anti-drug antibody (ADA) titer, of those who were ADA negative at baseline
Time Frame: Approximately 32 months
Population: For arms 0.0001 and 0.001 mg/kg of IV SL-279252, there were no subjects who were ADA negative at baseline. For arms 12.0 and 24.0 mg/kg of IV SL-279252, ADA samples were not collected.
Measure: Count of Participants; unit: Participants
Arm/Group | SL-279252 (0.0001 mg/kg S1) | SL-279252 (0.001 mg/kg S1) | SL-279252 (0.003 mg/kg S1) | SL-279252 (0.01 mg/kg S1) | SL-279252 (0.03 mg/kg S1) | SL-279252 (0.1 mg/kg S1) | SL-279252 (0.3 mg/kg S1) | SL-279252 (1.0 mg/kg S1) | SL-279252 (3.0 mg/kg S1) | SL-279252 (6.0 mg/kg S1) | SL-279252 (12.0 mg/kg S1) | SL-279252 (24.0 mg/kg S1) | SL-279252 (0.3 mg/kg S2) | SL-279252 (1.0 mg/kg S2) | SL-279252 (3.0 mg/kg S2)
Number analyzed (Participants) | 0 | 0 | 1 | 1 | 2 | 2 | 3 | 5 | 4 | 3 | 0 | 0 | 2 | 5 | 3
Participants | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 3 | 1 | 0 | 0 | 1 | 3 | 3

6. Secondary Outcome: Maximum Serum Concentration (Cmax) of SL-279252
Description: The Cmax is the maximum observed serum concentration of SL-279252 following single and multiple doses
Time Frame: Cycle 1 Day 1, Cycle 1 Day 15, and Cycle 2 Day 1 (cycle = 28 days)
Population: PK Population - number analyzed may be less than the number of participants in a given cohort if samples were not available for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- SL-279252 (0.3 mg/kg S1 or S2): 0.3 mg/kg of IV SL-279252 (Schedule 1 or Schedule 2)
- SL-279252 (1.0 mg/kg S1 or S2): 1.0 mg/kg of IV SL-279252 (Schedule 1 or Schedule 2)
- SL-279252 (3.0 mg/kg S1 or S2): 3.0 mg/kg of IV SL-279252 (Schedule 1 or Schedule 2)
Arm/Group | SL-279252 (0.0001 mg/kg S1) | SL-279252 (0.001 mg/kg S1) | SL-279252 (0.003 mg/kg S1) | SL-279252 (0.01 mg/kg S1) | SL-279252 (0.03 mg/kg S1) | SL-279252 (0.1 mg/kg S1) | SL-279252 (0.3 mg/kg S1 or S2) | SL-279252 (1.0 mg/kg S1 or S2) | SL-279252 (3.0 mg/kg S1 or S2) | SL-279252 (6.0 mg/kg S1) | SL-279252 (12.0 mg/kg S1) | SL-279252 (24.0 mg/kg S1)
Number analyzed (Participants) | 1 | 1 | 2 | 1 | 2 | 3 | 8 | 12 | 9 | 4 | 4 | 2
ng/mL
  Cycle 1 Day 1 | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | 3.75 (NA) — Geometric Coefficient of Variation not calculable for a single participant | 30.8 (4.60) | 93.4 (NA) — Geometric Coefficient of Variation not calculable for a single participant | 427 (1.82) | 734 (42.9) | 3580 (29.6) | 10200 (42.0) | 28100 (43.0) | 83600 (26.3) | 248000 (34.7) | 320000 (16.0)
  Cycle 1 Day 15: number analyzed (Participants) | 1 | 1 | 1 | 1 | 2 | 3 | 7 | 12 | 9 | 3 | 4 | 2
  Cycle 1 Day 15 | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | 3.22 (NA) — Geometric Coefficient of Variation not calculable for a single participant | 19.5 (NA) — Geometric Coefficient of Variation not calculable for a single participant | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | 360 (6.09) | 731 (35.9) | 2920 (52.9) | 10400 (45.9) | 26100 (67.0) | 75300 (21.5) | 277000 (10.5) | 349000 (4.05)
  Cycle 2 Day 1 (Schedule 1 only): number analyzed (Participants) | 1 | 1 | 2 | 0 | 2 | 3 | 4 | 5 | 5 | 2 | 4 | 2
  Cycle 2 Day 1 (Schedule 1 only) | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | 50.6 (49.2) |  | 408 (13.0) | 1090 (20.9) | 4260 (24.2) | 9760 (28.4) | 25400 (103) | 94100 (15.6) | 236000 (25.8) | 355000 (7.97)
  Cycle 2 Day 1 (Schedule 2 only): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 6 | 3 | 0 | 0 | 0
  Cycle 2 Day 1 (Schedule 2 only) |  |  |  |  |  |  | 4110 (13.4) | 11700 (36.9) | 38300 (22.7) |  |  |

7. Secondary Outcome: Minimum Serum Concentration (Cmin) of SL-279252
Description: The Cmin is the minimum observed serum concentration of SL-279252 following single and multiple doses
Time Frame: Cycle 1 Day 15 and Cycle 2 Day 1 (cycle = 28 days)
Population: PK Population - number analyzed may be less than the number of participants in a given cohort if samples were below the limit of quantitation or not available for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | SL-279252 (0.0001 mg/kg S1) | SL-279252 (0.001 mg/kg S1) | SL-279252 (0.003 mg/kg S1) | SL-279252 (0.01 mg/kg S1) | SL-279252 (0.03 mg/kg S1) | SL-279252 (0.1 mg/kg S1) | SL-279252 (0.3 mg/kg S1 or S2) | SL-279252 (1.0 mg/kg S1 or S2) | SL-279252 (3.0 mg/kg S1 or S2) | SL-279252 (6.0 mg/kg S1) | SL-279252 (12.0 mg/kg S1) | SL-279252 (24.0 mg/kg S1)
Number analyzed (Participants) | 1 | 1 | 2 | 1 | 2 | 3 | 7 | 12 | 9 | 3 | 4 | 1
ng/mL
  Cycle 1 Day 15 | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | 1.03 (71.9) | 3.77 (56.5) | 10.4 (124) | 29.0 (43.0) | 90.7 (100) | 12.7 (NA) — Geometric Coefficient of Variation not calculable for a single participant
  Cycle 2 Day 1 (Schedule 2 only): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 6 | 3 | 0 | 0 | 0
  Cycle 2 Day 1 (Schedule 2 only) |  |  |  |  |  |  | 1.12 (75.2) | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | 11.9 (164) |  |  |

8. Secondary Outcome: Time at Which Maximum Concentration of SL-279252 is Observed (Tmax)
Description: The Tmax is the time at which the maximum concentration of SL-279252 is observed following single and multiple doses
Time Frame: Cycle 1 Day 1, Cycle 1 Day 15, and Cycle 2 Day 1 (cycle = 28 days)
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | SL-279252 (0.0001 mg/kg S1) | SL-279252 (0.001 mg/kg S1) | SL-279252 (0.003 mg/kg S1) | SL-279252 (0.01 mg/kg S1) | SL-279252 (0.03 mg/kg S1) | SL-279252 (0.1 mg/kg S1) | SL-279252 (0.3 mg/kg S1 or S2) | SL-279252 (1.0 mg/kg S1 or S2) | SL-279252 (3.0 mg/kg S1 or S2) | SL-279252 (6.0 mg/kg S1) | SL-279252 (12.0 mg/kg S1) | SL-279252 (24.0 mg/kg S1)
Number analyzed (Participants) | 1 | 1 | 2 | 1 | 2 | 3 | 8 | 12 | 9 | 4 | 4 | 2
hours
  Cycle 1 Day 1 | NA [NA to NA] — Not estimable based on subjects' concentration profiles, including values below the limit of quantitation | 0.42 [0.42 to 0.42] | 1.89 [0.25 to 3.53] | 0.72 [0.72 to 0.72] | 0.78 [0.57 to 1.00] | 0.55 [0.53 to 0.67] | 0.53 [0.50 to 1.13] | 1.05 [0.58 to 1.52] | 1.05 [0.98 to 1.40] | 0.86 [0.58 to 1.07] | 1.40 [0.93 to 1.78] | 1.16 [1.02 to 1.30]
  Cycle 1 Day 15: number analyzed (Participants) | 1 | 1 | 1 | 1 | 2 | 3 | 7 | 12 | 9 | 3 | 4 | 2
  Cycle 1 Day 15 | NA [NA to NA] — Not estimable based on subjects' concentration profiles, including values below the limit of quantitation | 0.17 [0.17 to 0.17] | 0.33 [0.33 to 0.33] | NA [NA to NA] — Not estimable based on subjects' concentration profiles, including values below the limit of quantitation | 0.50 [0.50 to 0.50] | 0.50 [0.50 to 0.50] | 0.50 [0.50 to 0.50] | 1.00 [1.00 to 1.05] | 1.00 [1.00 to 3.00] | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.25] | 1.00 [1.00 to 1.00]
  Cycle 2 Day 1 (Schedule 1 only): number analyzed (Participants) | 1 | 1 | 2 | 0 | 2 | 3 | 4 | 5 | 5 | 2 | 4 | 2
  Cycle 2 Day 1 (Schedule 1 only) | NA [NA to NA] — Not estimable based on subjects' concentration profiles, including values below the limit of quantitation | NA [NA to NA] — Not estimable based on subjects' concentration profiles, including values below the limit of quantitation | 0.38 [0.27 to 0.50] |  | 0.55 [0.52 to 0.58] | 0.58 [0.53 to 0.60] | 0.54 [0.42 to 0.58] | 1.05 [0.58 to 1.38] | 1.38 [1.02 to 3.02] | 1.00 [0.95 to 1.05] | 1.17 [1.08 to 1.30] | 1.08 [1.05 to 1.12]
  Cycle 2 Day 1 (Schedule 2 only): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 6 | 3 | 0 | 0 | 0
  Cycle 2 Day 1 (Schedule 2 only) |  |  |  |  |  |  | 0.70 [0.53 to 0.88] | 1.04 [1.02 to 1.08] | 1.03 [1.03 to 1.03] |  |  |

9. Secondary Outcome: Area Under the Serum Concentration-time Curve (AUC)
Description: The AUC is the area under the serum concentration time curve following single and multiple doses of SL-279252. AUC (0-inf; from time 0 to infinity) is reported for C1D1 and C2D1 (Schedule 1 only); AUC (tau; over a dosing interval) is reported for C1D15 and C2D1 (Schedule 2 only).
Time Frame: Cycle 1 Day 1, Cycle 1 Day 15, and Cycle 2 Day 1 (cycle = 28 days)
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*ng/mL
Arm/Group | SL-279252 (0.0001 mg/kg S1) | SL-279252 (0.001 mg/kg S1) | SL-279252 (0.003 mg/kg S1) | SL-279252 (0.01 mg/kg S1) | SL-279252 (0.03 mg/kg S1) | SL-279252 (0.1 mg/kg S1) | SL-279252 (0.3 mg/kg S1 or S2) | SL-279252 (1.0 mg/kg S1 or S2) | SL-279252 (3.0 mg/kg S1 or S2) | SL-279252 (6.0 mg/kg S1) | SL-279252 (12.0 mg/kg S1) | SL-279252 (24.0 mg/kg S1)
Number analyzed (Participants) | 1 | 1 | 2 | 1 | 2 | 3 | 8 | 12 | 9 | 4 | 4 | 2
hours*ng/mL
  Cycle 1 Day 1 | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | 56.6 (77.5) | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | 804 (NA) — Geometric Coefficient of Variation not calculable for a single participant (one participant's concentrations were below limit of quantitation) | 2960 (40.1) | 10900 (39.2) | 38800 (32.7) | 110000 (52.9) | 353000 (29.4) | 1140000 (48.2) | 1380000 (22.4)
  Cycle 1 Day 15: number analyzed (Participants) | 1 | 1 | 1 | 1 | 2 | 3 | 7 | 12 | 9 | 3 | 4 | 2
  Cycle 1 Day 15 | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | 68.8 (NA) — Geometric Coefficient of Variation not calculable for a single participant | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | 3410 (47.4) | 11600 (43.5) | 40800 (38.9) | 130000 (40.5) | 325000 (31.5) | 1100000 (21.2) | 1390000 (16.9)
  Cycle 2 Day 1 (Schedule 1 only): number analyzed (Participants) | 1 | 1 | 2 | 0 | 2 | 3 | 4 | 5 | 5 | 2 | 4 | 2
  Cycle 2 Day 1 (Schedule 1 only) | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification |  | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | 3240 (35.7) | 10800 (43.7) | 36800 (24.1) | 103000 (15.3) | 388000 (28.2) | 1160000 (29.7) | 1560000 (15.0)
  Cycle 2 Day 1 (Schedule 2 only): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 6 | 3 | 0 | 0 | 0
  Cycle 2 Day 1 (Schedule 2 only) |  |  |  |  |  |  | 11500 (16.1) | 33600 (58.5) | 145000 (35.2) |  |  |

10. Secondary Outcome: Terminal Half Life (t1/2)
Description: The t1/2 elimination half-life of SL-279252
Time Frame: Cycle 1 Day 1, Cycle 1 Day 15, and Cycle 2 Day 1 (cycle = 28 days)
Population: PK Population - number analyzed may be less than the number of participants in a given cohort if samples were below the limit of quantitation or not available for analysis. Not estimable based on subjects' concentration profiles, including values below the limit of quantification
Measure: Median (Full Range); unit: hours
Arm/Group | SL-279252 (0.0001 mg/kg S1) | SL-279252 (0.001 mg/kg S1) | SL-279252 (0.003 mg/kg S1) | SL-279252 (0.01 mg/kg S1) | SL-279252 (0.03 mg/kg S1) | SL-279252 (0.1 mg/kg S1) | SL-279252 (0.3 mg/kg S1 or S2) | SL-279252 (1.0 mg/kg S1 or S2) | SL-279252 (3.0 mg/kg S1 or S2) | SL-279252 (6.0 mg/kg S1) | SL-279252 (12.0 mg/kg S1) | SL-279252 (24.0 mg/kg S1)
Number analyzed (Participants) | 1 | 1 | 2 | 1 | 2 | 3 | 8 | 12 | 9 | 4 | 4 | 2
hours
  Cycle 1 Day 1 | NA [NA to NA] — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | 2.69 [2.69 to 2.69] | 4.36 [2.23 to 6.49] | NA [NA to NA] — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | 1.23 [1.23 to 1.23] | 25.2 [2.49 to 26.3] | 23.4 [17.0 to 29.1] | 22.6 [15.3 to 24.9] | 22.4 [19.4 to 36.3] | 22.9 [19.1 to 27.3] | 20.0 [12.9 to 22.4] | 14.4 [10.5 to 18.3]
  Cycle 1 Day 15: number analyzed (Participants) | 1 | 1 | 1 | 1 | 2 | 3 | 7 | 12 | 9 | 3 | 4 | 2
  Cycle 1 Day 15 | NA [NA to NA] — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | NA [NA to NA] — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | 5.74 [5.74 to 5.74] | NA [NA to NA] — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | NA [NA to NA] — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | 5.30 [5.17 to 5.43] | 5.87 [4.86 to 6.95] | 6.00 [3.06 to 7.05] | 6.14 [5.34 to 7.01] | 6.48 [5.73 to 7.31] | 4.86 [4.82 to 5.60] | 4.13 [3.99 to 4.26]
  Cycle 2 Day 1 (Schedule 1 only): number analyzed (Participants) | 1 | 1 | 2 | 0 | 2 | 3 | 4 | 5 | 5 | 2 | 4 | 2
  Cycle 2 Day 1 (Schedule 1 only) | NA [NA to NA] — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | NA [NA to NA] — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | NA [NA to NA] — Not estimable based on subjects' concentration profiles, including values below the limit of quantification |  | NA [NA to NA] — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | 5.30 [3.10 to 5.51] | 5.22 [4.46 to 5.90] | 5.98 [5.70 to 6.56] | 5.48 [5.09 to 5.88] | 5.32 [4.64 to 6.00] | 4.71 [4.62 to 5.44] | 3.78 [3.34 to 4.23]
  Cycle 2 Day 1 (Schedule 2 only): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 6 | 3 | 0 | 0 | 0
  Cycle 2 Day 1 (Schedule 2 only) |  |  |  |  |  |  | 4.48 [4.31 to 5.50] | 5.09 [2.33 to 5.80] | 5.10 [4.18 to 5.79] |  |  |

11. Secondary Outcome: Clearance
Description: Clearance of SL-279252
Time Frame: Cycle 1 Day 1, Cycle 1 Day 15, and Cycle 2 Day 1 (cycle = 28 days)
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per hour per kg
Arm/Group | SL-279252 (0.0001 mg/kg S1) | SL-279252 (0.001 mg/kg S1) | SL-279252 (0.003 mg/kg S1) | SL-279252 (0.01 mg/kg S1) | SL-279252 (0.03 mg/kg S1) | SL-279252 (0.1 mg/kg S1) | SL-279252 (0.3 mg/kg S1 or S2) | SL-279252 (1.0 mg/kg S1 or S2) | SL-279252 (3.0 mg/kg S1 or S2) | SL-279252 (6.0 mg/kg S1) | SL-279252 (12.0 mg/kg S1) | SL-279252 (24.0 mg/kg S1)
Number analyzed (Participants) | 1 | 1 | 2 | 1 | 2 | 3 | 8 | 12 | 9 | 4 | 4 | 2
liters per hour per kg
  Cycle 1 Day 1 | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | 0.0530 (77.5) | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | 0.0373 (NA) — Geometric Coefficient of Variation not calculable for a single participant (one participant's concentrations were below limit of quantitation) | 0.0338 (40.1) | 0.0274 (39.2) | 0.0258 (32.7) | 0.0272 (52.9) | 0.0170 (29.4) | 0.0106 (48.2) | 0.0174 (22.4)
  Cycle 1 Day 15: number analyzed (Participants) | 1 | 1 | 1 | 1 | 2 | 3 | 7 | 12 | 9 | 3 | 4 | 2
  Cycle 1 Day 15 | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | 0.0436 (NA) — Geometric Coefficient of Variation not calculable for a single participant | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | 0.0293 (47.4) | 0.0258 (43.5) | 0.0245 (38.9) | 0.0231 (40.5) | 0.0184 (31.5) | 0.0109 (21.2) | 0.0172 (16.9)
  Cycle 2 Day 1 (Schedule 1 only): number analyzed (Participants) | 1 | 1 | 2 | 0 | 2 | 3 | 4 | 5 | 5 | 2 | 4 | 2
  Cycle 2 Day 1 (Schedule 1 only) | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification |  | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | 0.0309 (35.7) | 0.0277 (43.7) | 0.0272 (24.1) | 0.0291 (15.3) | 0.0155 (28.2) | 0.0103 (29.7) | 0.0154 (15.0)
  Cycle 2 Day 1 (Schedule 2 only): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 6 | 3 | 0 | 0 | 0
  Cycle 2 Day 1 (Schedule 2 only) |  |  |  |  |  |  | 0.0261 (16.1) | 0.0298 (58.5) | 0.0207 (35.2) |  |  |

12. Secondary Outcome: Volume of Distribution
Description: Volume of distribution of SL-279252
Time Frame: Cycle 1 Day 1, Cycle 1 Day 15, and Cycle 2 Day 1 (cycle = 28 days)
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per kg
Arm/Group | SL-279252 (0.0001 mg/kg S1) | SL-279252 (0.001 mg/kg S1) | SL-279252 (0.003 mg/kg S1) | SL-279252 (0.01 mg/kg S1) | SL-279252 (0.03 mg/kg S1) | SL-279252 (0.1 mg/kg S1) | SL-279252 (0.3 mg/kg S1 or S2) | SL-279252 (1.0 mg/kg S1 or S2) | SL-279252 (3.0 mg/kg S1 or S2) | SL-279252 (6.0 mg/kg S1) | SL-279252 (12.0 mg/kg S1) | SL-279252 (24.0 mg/kg S1)
Number analyzed (Participants) | 1 | 1 | 2 | 1 | 2 | 3 | 8 | 12 | 9 | 4 | 4 | 2
liters per kg
  Cycle 1 Day 1 | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | 0.291 (6.92) | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | 0.0664 (NA) — Geometric Coefficient of Variation not calculable for a single participant (one participant's concentrations were below limit of quantitation) | 0.576 (144) | 0.894 (38.0) | 0.797 (31.8) | 0.939 (52.8) | 0.562 (33.8) | 0.281 (64.8) | 0.348 (17.4)
  Cycle 2 Day 1 (Schedule 1 only): number analyzed (Participants) | 1 | 1 | 2 | 0 | 2 | 3 | 4 | 5 | 5 | 2 | 4 | 2
  Cycle 2 Day 1 (Schedule 1 only) | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification |  | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantification | 0.200 (46.3) | 0.207 (37.1) | 0.237 (23.7) | 0.229 (12.5) | 0.118 (9.5) | 0.0730 (20.5) | 0.0834 (32.3)
  Cycle 2 Day 1 (Schedule 2 only): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 6 | 3 | 0 | 0 | 0
  Cycle 2 Day 1 (Schedule 2 only) |  |  |  |  |  |  | 0.178 (8.63) | 0.189 (30.4) | 0.149 (47.1) |  |  |

ADVERSE EVENTS:
Time Frame: Subjects were followed continuously for all AEs starting when a subject signed the informed consent form, throughout the course of treatment, and for 90 days after the last dose of study treatment, an average of 17 weeks.
Arm/Group | SL-279252 (0.0001 mg/kg S1) | SL-279252 (0.001 mg/kg S1) | SL-279252 (0.003 mg/kg S1) | SL-279252 (0.01 mg/kg S1) | SL-279252 (0.03 mg/kg S1) | SL-279252 (0.1 mg/kg S1) | SL-279252 (0.3 mg/kg S1) | SL-279252 (1.0 mg/kg S1) | SL-279252 (3.0 mg/kg S1) | SL-279252 (6.0 mg/kg S1) | SL-279252 (12.0 mg/kg S1) | SL-279252 (24.0 mg/kg S1) | SL-279252 (0.3 mg/kg S2) | SL-279252 (1.0 mg/kg S2) | SL-279252 (3.0 mg/kg S2)
All-Cause Mortality (participants affected / at risk) | 1/1 | 1/1 | 2/2 | 1/1 | 0/2 | 3/3 | 4/4 | 4/6 | 5/6 | 4/4 | 2/4 | 0/2 | 2/4 | 5/6 | 3/3
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/1 | 0/2 | 0/1 | 0/2 | 1/3 | 1/4 | 3/6 | 1/6 | 1/4 | 0/4 | 1/2 | 0/4 | 2/6 | 1/3
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 2/2 | 1/1 | 2/2 | 3/3 | 4/4 | 4/6 | 6/6 | 3/4 | 4/4 | 2/2 | 4/4 | 5/6 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SL-279252 (0.0001 mg/kg S1) (N=1) | SL-279252 (0.001 mg/kg S1) (N=1) | SL-279252 (0.003 mg/kg S1) (N=2) | SL-279252 (0.01 mg/kg S1) (N=1) | SL-279252 (0.03 mg/kg S1) (N=2) | SL-279252 (0.1 mg/kg S1) (N=3) | SL-279252 (0.3 mg/kg S1) (N=4) | SL-279252 (1.0 mg/kg S1) (N=6) | SL-279252 (3.0 mg/kg S1) (N=6) | SL-279252 (6.0 mg/kg S1) (N=4) | SL-279252 (12.0 mg/kg S1) (N=4) | SL-279252 (24.0 mg/kg S1) (N=2) | SL-279252 (0.3 mg/kg S2) (N=4) | SL-279252 (1.0 mg/kg S2) (N=6) | SL-279252 (3.0 mg/kg S2) (N=3)
acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
inguinal hernia, obstructive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SL-279252 (0.0001 mg/kg S1) (N=1) | SL-279252 (0.001 mg/kg S1) (N=1) | SL-279252 (0.003 mg/kg S1) (N=2) | SL-279252 (0.01 mg/kg S1) (N=1) | SL-279252 (0.03 mg/kg S1) (N=2) | SL-279252 (0.1 mg/kg S1) (N=3) | SL-279252 (0.3 mg/kg S1) (N=4) | SL-279252 (1.0 mg/kg S1) (N=6) | SL-279252 (3.0 mg/kg S1) (N=6) | SL-279252 (6.0 mg/kg S1) (N=4) | SL-279252 (12.0 mg/kg S1) (N=4) | SL-279252 (24.0 mg/kg S1) (N=2) | SL-279252 (0.3 mg/kg S2) (N=4) | SL-279252 (1.0 mg/kg S2) (N=6) | SL-279252 (3.0 mg/kg S2) (N=3)
constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 3 | 1
decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 1 | 1
back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 1 | 1 | 0 | 1 | 0 | 0
infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 1 | 2
anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 2 | 1
insomnia (Psychiatric disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 2 | 1
cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0
rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1
dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1
headache (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0
neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
face oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
localised oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
sacral pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
anosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
rhonci (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
thoracic haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
corneal abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
blood iron decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
breast pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
eyelid function disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
blood creatine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site agrees not to publish any Study Results or data before the publication of results from the Overall Study. After Sponsor has published the results of the Overall Study, Site may publish or present results generated at Site. If Sponsor has not published results of the Overall Study within 18 months of data base lock, Site may publish the results of the Study that were generated at Site. Site agrees to first submit to Sponsor the proposed publication at least 30 days prior to the submission.

DOCUMENTS (2):
  • Study Protocol (2021-07-12): https://cdn.clinicaltrials.gov/large-docs/18/NCT03894618/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-04): https://cdn.clinicaltrials.gov/large-docs/18/NCT03894618/SAP_001.pdf